CLINICAL TRIAL: NCT05878847
Title: Oral Supplement in Older Adults to Support Physical Fitness and Mental Well-being
Acronym: PQQA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aberystwyth University (Other)
Collaborators: Phytoquest Ltd (Unknown); Gateway Health Alliances, Inc (Unknown); Welsh Government (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 23767; PQQA (Other: WARU)
Record Dates: First submitted 2023-04-20; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-04

CONDITIONS: Osteo-arthritis
Keywords: Older adults; Mental well-being; Physical fitness; Sleep quality
MeSH Terms: conditions — Psychological Well-Being; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study is split into three experimental sessions where you will be randomised to one of two supplements, Q-actin (2 x 10 mg gummies daily) or placebo (2 x 10 mg gummies daily) supplementation for 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Q-actin (Experimental): Q-actin gummies (2 x 10mg) daily for 12 weeks
  Interventions: Dietary Supplement: Q-actin
- Placebo (Placebo Comparator): Placebo gummies (2 x 10mg) daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Q-actin — idoBR1 is an iminosugar amino acid isolated from fruits of certain cucumbers, Cucumis sativus (Cucurbitaceae), which has been shown to have anti-inflammatory activity. IminoTech Inc in the USA has produced a quality-controlled cucumber extract containing measured idoBR1 (Q-actin™) that has given good results in osteo-arthritis from oral use.
  Other Names: idoBR1
  Arms: Q-actin
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Cucumbers have been anecdotally claimed to have anti-inflammatory activity for a long time, but the active principle was not identified. idoBR1 is an iminosugar amino acid isolated from fruits of certain cucumbers, Cucumis sativus (Cucurbitaceae), which has been shown to have anti-inflammatory activity. IminoTech Inc in the USA has produced a quality-controlled cucumber extract containing measured idoBR1 (Q-actin™) that has given good results in osteo-arthritis from oral use.

The investigators are aiming to recruit a cohort (n = 50) of middle aged and older adults (>50 years) who will be randomised into Q-actin (2 x 10 mg gummies daily) or placebo (2 x 10 mg gummies daily) supplementation for 12 weeks. Using hand grip strength and the Nine-Hole Peg Test (9HPT) the investigators will measure physical strength and finger dexterity respectively. The investigators will measure generic quality of life with the EuroQol 5 Dimension 5 (EQ-5D) questionnaire, sleep quality, diet choices and collect urine samples for the investigation into the chemical composition (metabolomics).

Randomisation will be blinded, and the participant and the researcher will not know what group participants in until after the completion of the study, then it will be disclosed.

DETAILED DESCRIPTION:
Cucumbers have been anecdotally claimed to have anti-inflammatory activity for a long time, but the active principle was not identified. idoBR1 is an iminosugar amino acid isolated from fruits of certain cucumbers, Cucumis sativus (Cucurbitaceae), which has been shown to have anti-inflammatory activity.

The investigators would like to explore if consumption of cucumber extract Q-actin when compared with placebo can have an impact on physical strength (measured by hand grip strength), finger dexterity (measured by Nine-Hole Peg Test (9HPT)) as well as quality of life (EuroQol 5 Dimension 5: EQ-5D questionnaire), sleep quality (Pittsburgh Sleep Quality Index), and diet (diet questionnaires are tailored to the participants eating habits, e.g., carnivore, vegetarian, fish, vegan etc). The investigators will explore urine chemical composition use high resolution metabolomics do this by looking at the chemical composition of home-collected urine.

After pre-induction over the phone, if the person is eligible and still interested, the investigators will firstly run through an induction session. This can be done by phone, Teams or in person, whatever suits best. The study is split into three experimental sessions where the participant will be randomised to one of two supplements, Q-actin (2 x 10 mg gummies daily) or placebo (2 x 10 mg gummies daily) supplementation for 12 weeks. The vegan gummies will need to be consumed in the evening, before bed-time. Randomisation will be blinded, and the participant and the researcher will not know what group they in until after the completion of the study. The participant will need to come to the centre for physical strength and finger dexterity measurements using hand grip strength and the Nine-Hole Peg Test (9HPT) respectively. The investigators will measure generic quality of life with the EQ-5D questionnaire, record diet choices, record sleeping habits using the Pittsburgh Sleep Quality Index, and collect urine samples before and after the supplementation period. The investigators would like participants to restrict from consumption of cucumber, gherkins, and melon for two days before coming to the centre.

Whilst undergoing the study, if necessary, the research team will be easily contacted by email, Teams and phone.

The visits

Tea, coffee and biscuits will be provided at each visit. Each visit will take up to an hour

Induction

First, the participant will be welcomed with tea or coffee. The investigators will run through how the investigators are working safely during coronavirus (COVID-19). Then the investigators will introduce the participant to the urine sampling boxes, provide crib sheets and email the participant with a link to a video demonstration, if needed. The investigators will run through the logistics of study visits and the tasks that will be completed.

The investigators will also email the participant a link to the EQ-5D questionnaire, Pittsburgh Sleep Quality Index, and diet questionnaire, or give them a paper copy, so that they can complete these in the centre or at home (whatever is preferred).

The investigators will arrange the participants testing day 1, 2 and 3 visit dates and times.

Testing day 1 (start)

On the participants pre-organised day and time, will will ask them to collect 2 x 4ml first urine sample at home using home-collection urine kits. These samples will be stored in the participants home home fridge between 2-5 degrees. The participant will then come to the centre at a pre-organised timeslot with their urine samples for physical strength and finger dexterity activities. Will will ask them to make sure they complete their EQ-5D, Pittsburgh Sleep Quality Index, and diet questionnaire before they start their supplementation.

Testing day 2 (after 6 weeks)

After the 6-week supplementation period the investigators would like the participant to complete the activities that they undertook during testing day 1.

On their pre-organised day and time, will will ask them to collect 2 x 4ml first urine sample at home using home-collection urine kits. The investigators will ask the participant to store these samples in their home fridge between 2-5 degrees. The participant will then come to the centre for their pre-organised timeslot with their urine samples for physical strength and finger dexterity activities. The investigators will ask the participant to make sure they complete their EQ-5D, Pittsburgh Sleep Quality index, and diet questionnaire before or just after testing day 2.

Testing day 3 (after 12 weeks)

After the 12-week supplementation period the investigators would like the participant to complete the activities that they undertook during testing day 1.

On their pre-organised day and time, will will ask them to collect 2 x 4ml first urine sample at home using home-collection urine kits. The investigators will ask the participant to store these samples in their home fridge between 2-5 degrees. The participant will then come to the centre for their pre-organised timeslot with their urine samples for physical strength and finger dexterity activities. The investigators will ask the participant to make sure they complete their EQ-5D, Pittsburgh Sleep Quality index, and diet questionnaire before or just after testing day 3.

There will also be an optional feedback questionnaire at the end.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years, mixed gender, mixed ethnicity
* Consenting adults >50 y Age
* Commit to urine sampling
* Able to commit to attending WARU or the remote centre for measurements of physical strength, finger dexterity, quality of life, diet choices, sleep Able to restrict from consumption of cucumber, gherkins, and melon for two days before coming to WARU or the remote centre

Exclusion Criteria:

* Showing (or anyone within the household) any COVID-19 symptoms (see COVID-19 basic health screen)*
* Higher risk or vulnerable from coronavirus or live with someone at a higher risk of a severe illness from COVID-19 (over 70, undergoing cancer treatment, high risk of getting infections).
* Had a letter from the NHS advising you to shield (isolate)
* Had been at risk of exposure to COVID-19 such as travel, contact with someone with COVID-19, been exposed to the virus, or has been asked to self-isolate by the track and trace system.
* Serious health conditions that require daily long-term medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Physical strength | Change from Baseline grip strength at 12 weeks
  Hand grip strength using a hand held dynamometer
Finger dexterity measurements | Change from baseline Finger dexterity at 12 weeks
  Nine-Hole Peg Test (9HPT)

SECONDARY OUTCOMES:
EuroQol 5 Dimension 5L (combined score) | Reduced score from baseline EuroQol 5 Dimension 5 score at 12 weeks.
  EuroQol 5 Dimension 5 5L questionnaire: Generic quality of life. Mobility- Level 1-5 Self-Care- Level 1-5, Usual Activities- Level 1-5, Pain/Discomfort- Level 1-5, Anxiety/Depression- Level 1-5. The digits for the five dimensions will be combined into a 5-digit number that describes the patient's health state.
Diet choices | Increased score from baseline Prime Diet Quality Score at 12 weeks
  Measured using the Prime Diet Quality Score. The PDQS measures intake of the 22 component foods/food groups over the last 30 days with seven possible responses for each component ranging from "once a month or less" to "≥ 2 times/day." Scores are then summed to create a PDQS total diet quality score with a possible score from 0 to 126 with higher scores indicating a healthier diet.
Record sleeping habits | Decreased score from baseline Pittsburgh Sleep Quality Index at 12 weeks
  Pittsburgh Sleep Quality Index Component 1: Subjective sleep quality-question 9 Component 2: Sleep latency-questions 2 and 5a Component 3: Sleep duration-question 4 Component 4: Sleep efficiency-questions 1, 3, and 4 Component 5: Sleep disturbance-questions 5b-5j Component 6: Use of sleep medication-question 6 Component 7: Daytime dysfunction-questions 7 and 8 Global PSQI Score: Sum of seven component scores

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Jane J Lloyd, PhD, BSc, Principal Investigator — Aberystwyth University
Locations (1):
- Well-being and Health Assessment Research Unit (WARU), Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be made available to other researchers.

REFERENCES:
- [Derived] Lloyd AJ, Nash RJ, Warren-Walker A, Watson A, Martinez Martin MP, Davies C, Villarreal-Ramos B, Wilson T, Beckmann M. Oral supplement in healthy older adults to support physical fitness and mental wellbeing. Front Nutr. 2025 May 12;12:1563999. doi: 10.3389/fnut.2025.1563999. eCollection 2025. PMID 40421033

DOCUMENTS (1):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05878847/Prot_000.pdf